CLINICAL TRIAL: NCT04286568
Title: Wald Outreach for Wellness
Brief Title: Wald Outreach for Wellness: Blood Pressure Outreach
Acronym: WOW
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Disruption by Covid-19.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00243167
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-08

CONDITIONS: Pre-hypertension; Hypertension
Keywords: Health Disparities; Outreach; Health Behavior; Under-served communities
MeSH Terms: conditions — Prehypertension; Hypertension; Health Behavior

STUDY DESIGN:
Intervention Model Description: quasi-experimental non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WOW Intervention (Experimental): Participants will receive blood pressure monitor and health passport to record blood pressure readings for 3 months.
  Participants will receive daily text message reminders to take and record blood pressure readings.
  Participants will receive health education and health care navigation. Participants will be assessed for social determinants of health. Participants will take surveys 3 times over 3 months. Participants will receive home visits or phone calls to collect data and receive health coaching.
  Interventions: Behavioral: WOW Intervention

INTERVENTIONS:
Behavioral: WOW Intervention — Health education and coaching, health care navigation,

SUMMARY:
The Wald Outreach Center will partner with Medicine for the Greater Good (MGG) to implement this pilot project called Wald Outreach for Wellness (WOW), a blood pressure outreach wellness intervention in a retail setting.

DETAILED DESCRIPTION:
WOW aims to provide community members with a digital blood pressure monitor, health education, and health care navigation as practical strategies to improve community members' management of pre-hypertension, and to reduce associated burdens and risks related to hypertension health disparities.

This approach to reaching populations who use retail settings has the potential to implement a health promotion and wellness strategy aimed at populations with increased risk for hypertension related health disparities. The outreach strategy is aimed at reaching community members where community members gather for health care, provide the community members with practical, low-cost strategies for promoting health and wellness, increase community members' knowledge in hypertension management, help the community members navigate health care options and get the community members engaged in a medical home thereby reducing the burdens of hypertension health disparities.

This research is important to continue to assess the best ways to reach and reduce hypertension health disparities in underserved communities with limited access to health care.

ELIGIBILITY:
Inclusion Criteria:

* Community residents who participate in Day at the Market
* Adult individuals 18 years and older whose recorded BP reading is within the pre-hypertensive range 120-139 systolic; 80-89 diastolic
* Able to read and understand English

Exclusion Criteria:

* 17 years or younger
* BP reading above pre-hypertensive range
* Unable to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change in actions to control hypertension as assessed by the Behavioral Risk Factor Surveillance System Module 7 | Assessed at baseline, 6 weeks and 12 weeks
  Change in yes/no answers assessed by Behavioral Risk Factor Surveillance System (BRFSS) Module 7. 10 questions graded by yes/no response.
Change in blood pressure | Assessed at baseline and every 2 weeks, up to 3 months
  Change in blood pressure (BP) measured in mmHg.

SECONDARY OUTCOMES:
Change in usage of BP monitor | Assessed at baseline and every 2 weeks, up to 3 months
  Change in usage of blood pressure monitor assessed by number of BP readings done by participants.
Change in knowledge of the signs and symptoms of a heart attack and stroke as assessed by BRFSS Module 8 | Assessed at baseline, 6 weeks and 12 weeks
  Change in knowledge (yes/no responses) of signs and symptoms of stroke/heart attack as assessed by BRFSS Module 8. 13 Questions graded by yes/no.
Change in engagement with healthcare provider as assessed by BRFSS Section 3 | Assessed at baseline, 6 weeks and 12 weeks
  Change in engagement with healthcare provider/medical home as assessed by BRFSS Section 3. 3 questions graded by yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ling, PhD, FNP-BC, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins University School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No